CLINICAL TRIAL: NCT02017756
Title: A Phase II Study of Chinese Atherosclerosis Risk Evaluation: Investigation of Carotid Atherosclerotic Disease in Patients With Ischemic Cerebrovascular Events
Brief Title: Chinese Atherosclerosis Risk Evaluation- Phase II
Acronym: CARE-II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Chun Yuan, Professor, Tsinghua University
Other Study IDs: Tsinghua-985
Record Dates: First submitted 2013-12-04; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack; Carotid Atherosclerotic Disease
Keywords: Carotid artery; Atherosclerosis; Vulnerable plaque; Magnetic resonance imaging; Arterial wall
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Carotid Artery Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Stroke is the first and the fourth leading cause of death in the United States and China, respectively. Disruption of cerebrovascular vulnerable atherosclerotic plaque is the major etiology of ischemic stroke. Therefore, early detection and treatment of vulnerable plaques occurring at the feeding arteries to brain (cerebral arteries) will be helpful for prevention of stroke.

Atherosclerosis is a systemic disease that usually affects multiple vascular beds. Previous studies have shown that these high risk lesions in different segments of cerebral arteries (intracranial and extracranial arteries) might be racially specific. It is reported that, in stroke patients, intracranial vulnerable plaques are prevalent in Asian populations whereas atherosclerosis more frequently involves extracranial carotid arteries in American subjects. However, these findings are based on angiographic imaging approaches via measuring arterial luminal stenosis. Because the atherosclerotic plaque often appears as outward expansion, namely positive remodeling during progression, measuring luminal stenosis will underestimate the disease severity. Hence, directly viewing the plaque in the vessel wall is strongly suggested in order to objectively evaluate the cerebrovascular vulnerable plaque.

High resolution, black-blood magnetic resonance (MR) imaging has been widely used to accurately characterize carotid vulnerable plaque in the last two decades. The aim of using MR black-blood techniques is to suppress the blood signal (black) to enhance the signal contrast between the vessel wall and blood in the arterial lumen. Excellent agreement has been achieved between MR imaging and histology in identification of plaque components, such as intraplaque hemorrhage and lipid core. For assessing carotid plaque, MR imaging is superior to computed tomography and ultrasound imaging techniques due to its advantages including noninvasive imaging, lack of ionizing radiation, excellent soft tissue resolution, and multi-parametric image acquisition.

The Investigators hypothesize that there are specific characteristics in carotid vulnerable plaques in Chinese patients with ischemic cerebrovascular events such as ischemic stroke and transient ischemic attack (TIA). This study seeks to investigate the characteristics of vulnerable plaque in carotid arteries using high resolution, black-blood MR imaging in patients with recent TIA or ischemic stroke.

This is a cross-sectional, multicenter study. A total of 1000 patients will be recruited from more than 10 different hospitals across China within 3 years. All patients will undergo MR imaging for brain and carotid arteries within two weeks after symptom onset. The prevalence of carotid vulnerable plaque and its correlations with brain ischemic lesions, traditional risk factors, and regional distribution of China will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent TIA of ischemic stroke (2 weeks) and carotid plaque determined by ultrasound will be included in this study.

Exclusion Criteria:

* Patients with contraindications to MR scan
* Patients with hemorrhagic stroke
* Patients with evidence of cardiogenic stroke
* Patients with brain tumors
* Patients underwent carotid revascularization therapy, such as stenting and endarterectomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, we plan to recruit patients with recent TIA of ischemic stroke (within 2 weeks) and carotid atherosclerotic plaque determined by ultrasound. The patients will be recruited from more than 10 hospitals in different areas of China.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of carotid vulnerable plaques, defined as lesions with intraplaque hemorrhage, fibrous cap rupture, or lipid core occupying >40% of vessel wall area as determined by high resolution, black-blood MR imaging in this study population. | within two weeks after symptom onset

SECONDARY OUTCOMES:
Carotid wall and brain infarct measurements. | within two weeks after symptom onset
  The following features will be measured: carotid mean wall thickness, normalized wall index, and incidence of compositional features (calcification, lipid core, intraplaque hemorrhage, cap rupture) and volume of cerebral white matter lesions or infarcts.
  These measurements will be used to determine the relationship of carotid wall features with the volume of cerebral white matter lesions or infarcts.
Traditional risk factors. | within two weeks after symptom onset
  Traditional risk factors will be collected from subjects including: age, gender, hypertension, smoke, diabetes, and history of cardiovascular disease. The association of the volume and incidence of carotid plaque calcification, lipid core, and intraplaque hemorrhage with traditional risk factors will be evaluated.
Incidence and volume of carotid plaques and geographic region of subjects. | within two weeks after symptom onset
  The incidence and the volume of carotid plaque calcification, lipid core, and intraplaque hemorrhage will be measured and collected. Data on geographic region of subjects in China, such as Northeast, North, East, South, and Western areas will be collected. This data will be used to study compare incidence and volume of carotid plaque features with geographic regions of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Yuan, PhD, Principal Investigator — Center for Biomedical Imaging Research, Department of Biomedical Engineering, Tsinghua University
Locations (14):
- China (14):
  - Department of Radiology, Peking University First Hospital, Beijing
  - Center for Biomedical Imaging Research, Department of Biomedical Engineering, Tsinghua University, Beijing
  - Department of Radiology, Beijing Hospital, Beijing
  - Department of Radiology, PLA General Hospital, Beijing
  - Department of Radiology, Fujian Medical University Union Hospital, Fuzhou
  - Department of Radiology, Sun Yat-Sen Memorial Hospital, Guangzhou
  - Department of Radiology, Zhujiang Hospital of Southern Medical University, Guangzhou
  - Department of Radiology, Harbin University The Fourth Affiliated Hospital, Harbin
  - Shandong Medical Imaging Research Institute, Jinan
  - Department of Radiology, Nanjing Drum Tower Hospital, Nanjing
  - Department of Radiology, The First Hospital of Qiqihaer City, Qiqihar
  - Department of Radiology, Shanghai Renji Hospital, Shanghai
  - Department of Radiology, Tianjin Fourth Centre Hospital, Tianjin
  - Department of Radiology, Qinghai University Affiliated Hospital, Xining

REFERENCES:
- [Background] Liu L, Wang D, Wong KS, Wang Y. Stroke and stroke care in China: huge burden, significant workload, and a national priority. Stroke. 2011 Dec;42(12):3651-4. doi: 10.1161/STROKEAHA.111.635755. Epub 2011 Nov 3. PMID 22052510
- [Background] Wong KS, Li H, Chan YL, Ahuja A, Lam WW, Wong A, Kay R. Use of transcranial Doppler ultrasound to predict outcome in patients with intracranial large-artery occlusive disease. Stroke. 2000 Nov;31(11):2641-7. doi: 10.1161/01.str.31.11.2641. PMID 11062288
- [Background] Saam T, Underhill HR, Chu B, Takaya N, Cai J, Polissar NL, Yuan C, Hatsukami TS. Prevalence of American Heart Association type VI carotid atherosclerotic lesions identified by magnetic resonance imaging for different levels of stenosis as measured by duplex ultrasound. J Am Coll Cardiol. 2008 Mar 11;51(10):1014-21. doi: 10.1016/j.jacc.2007.10.054. PMID 18325441
- [Background] Glagov S, Weisenberg E, Zarins CK, Stankunavicius R, Kolettis GJ. Compensatory enlargement of human atherosclerotic coronary arteries. N Engl J Med. 1987 May 28;316(22):1371-5. doi: 10.1056/NEJM198705283162204. PMID 3574413
- [Background] Cai JM, Hatsukami TS, Ferguson MS, Small R, Polissar NL, Yuan C. Classification of human carotid atherosclerotic lesions with in vivo multicontrast magnetic resonance imaging. Circulation. 2002 Sep 10;106(11):1368-73. doi: 10.1161/01.cir.0000028591.44554.f9. PMID 12221054
- [Background] Yuan C, Mitsumori LM, Ferguson MS, Polissar NL, Echelard D, Ortiz G, Small R, Davies JW, Kerwin WS, Hatsukami TS. In vivo accuracy of multispectral magnetic resonance imaging for identifying lipid-rich necrotic cores and intraplaque hemorrhage in advanced human carotid plaques. Circulation. 2001 Oct 23;104(17):2051-6. doi: 10.1161/hc4201.097839. PMID 11673345
- [Background] Saam T, Cai JM, Cai YQ, An NY, Kampschulte A, Xu D, Kerwin WS, Takaya N, Polissar NL, Hatsukami TS, Yuan C. Carotid plaque composition differs between ethno-racial groups: an MRI pilot study comparing mainland Chinese and American Caucasian patients. Arterioscler Thromb Vasc Biol. 2005 Mar;25(3):611-6. doi: 10.1161/01.ATV.0000155965.54679.79. Epub 2005 Jan 13. PMID 15653565
- [Derived] Shao S, Sun Y, Shi H, Li R, Sun Q, Yao B, Watase H, Hippe DS, Yuan C, Wang G, Zhang Q, Zhao X; Investigators of CARE-II Study. Metabolically Abnormal Obesity and Carotid Plaque Vulnerability: A Vessel Wall MRI Study Linking Obesity Phenotypes to Atherosclerotic Instability. Arterioscler Thromb Vasc Biol. 2025 Nov;45(11):2097-2108. doi: 10.1161/ATVBAHA.125.323413. Epub 2025 Sep 18. PMID 40964717
- [Derived] Meddings Z, Rundo L, Sadat U, Zhao X, Teng Z, Graves MJ. Robustness and classification capabilities of MRI radiomic features in identifying carotid plaque vulnerability. Br J Radiol. 2024 May 29;97(1158):1118-1124. doi: 10.1093/bjr/tqae057. PMID 38711198
- [Derived] Shao S, Shi H, Wang G, Li R, Sun Q, Yao B, Watase H, Hippe DS, Yuan C, Zhao X; Investigators of CARE-II study. Differences in left and right carotid plaque vulnerability in patients with bilateral carotid plaques: a CARE-II study. Stroke Vasc Neurol. 2023 Aug;8(4):284-291. doi: 10.1136/svn-2022-001937. Epub 2023 Jan 3. PMID 36596656
- [Derived] Baylam Geleri D, Watase H, Chu B, Chen L, Zhao H, Zhao X, Hatsukami TS, Yuan C; CARE-II Study Collaborators. Detection of Advanced Lesions of Atherosclerosis in Carotid Arteries Using 3-Dimensional Motion-Sensitized Driven-Equilibrium Prepared Rapid Gradient Echo (3D-MERGE) Magnetic Resonance Imaging as a Screening Tool. Stroke. 2022 Jan;53(1):194-200. doi: 10.1161/STROKEAHA.120.032505. Epub 2021 Sep 30. PMID 34587796
- [Derived] Jiang C, Zhang J, Zhu J, Wang X, Wen Z, Zhao X, Yuan C; CARE-II Investigators. Association between coexisting intracranial artery and extracranial carotid artery atherosclerotic diseases and ipsilateral cerebral infarction: a Chinese Atherosclerosis Risk Evaluation (CARE-II) study. Stroke Vasc Neurol. 2021 Dec;6(4):595-602. doi: 10.1136/svn-2020-000538. Epub 2021 Apr 26. PMID 33903178
- [Derived] Yang D, Ji Y, Wang D, Watase H, Hippe DS, Zhao X, Yuan C. Comparison of carotid atherosclerotic plaques between subjects in Northern and Southern China: a Chinese atherosclerosis risk evaluation study. Stroke Vasc Neurol. 2020 Jun;5(2):138-145. doi: 10.1136/svn-2019-000288. Epub 2020 Jan 29. PMID 32404502
- [Derived] Liu Y, Wang M, Zhang B, Wang W, Xu Y, Han Y, Yuan C, Zhao X. Size of carotid artery intraplaque hemorrhage and acute ischemic stroke: a cardiovascular magnetic resonance Chinese atherosclerosis risk evaluation study. J Cardiovasc Magn Reson. 2019 Jul 1;21(1):36. doi: 10.1186/s12968-019-0548-1. PMID 31262337
- [Derived] Zhou C, Yuan C, Li R, Wang W, Li C, Zhao X; CARE-II Study Collaborators. Association Between Incomplete Circle of Willis and Carotid Vulnerable Atherosclerotic Plaques. Arterioscler Thromb Vasc Biol. 2018 Nov;38(11):2744-2749. doi: 10.1161/ATVBAHA.118.311797. PMID 30354232
- [Derived] Zhao X, Li R, Hippe DS, Hatsukami TS, Yuan C; CARE-II Investigators. Chinese Atherosclerosis Risk Evaluation (CARE II) study: a novel cross-sectional, multicentre study of the prevalence of high-risk atherosclerotic carotid plaque in Chinese patients with ischaemic cerebrovascular events-design and rationale. Stroke Vasc Neurol. 2017 Feb 24;2(1):15-20. doi: 10.1136/svn-2016-000053. eCollection 2017 Mar. PMID 28959486
- [Derived] Zhao X, Hippe DS, Li R, Canton GM, Sui B, Song Y, Li F, Xue Y, Sun J, Yamada K, Hatsukami TS, Xu D, Wang M, Yuan C; CARE-II Study Collaborators. Prevalence and Characteristics of Carotid Artery High-Risk Atherosclerotic Plaques in Chinese Patients With Cerebrovascular Symptoms: A Chinese Atherosclerosis Risk Evaluation II Study. J Am Heart Assoc. 2017 Aug 14;6(8):e005831. doi: 10.1161/JAHA.117.005831. PMID 28862936